CLINICAL TRIAL: NCT01057719
Title: Climate Influence on Physiotherapy in Multiple Sclerosis
Acronym: CIOPIMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Oslo University Hospital (Other); University Hospital, Akershus (Other); University of Bergen (Other)
Responsible Party: Tori Smedal, Haukeland University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 012.06
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2010-01

CONDITIONS: Multiple Sclerosis
Keywords: cross-over design; mixed model; multiple sclerosis; physical performance measures; physical therapy; the Bobath concept; warm climate; 6-minute walk test
MeSH Terms: conditions — Multiple Sclerosis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiotherapy in Spain (Experimental): Daily inpatient physiotherapy for four weeks in a warm climate
  Interventions: Other: Physiotherapy
- Physiotherapy in Norway (Experimental): Daily inpatient physiotherapy for four weeks in a cold climate
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — Individual tailored physiotherapy according to the Bobath concept sixty minutes each working day for four weeks
  Other Names: Physical Therapy; Subtropical climate

SUMMARY:
The aim of the study was to compare the effect of inpatient physiotherapy in a warm climate versus physiotherapy in a colder climate in multiple sclerosis (MS), in both short- and long term perspectives.

DETAILED DESCRIPTION:
Empirically, several patients with MS have reported improved function in warm climate during therapy or vacation. This is in contrast to the heat intolerance frequently reported in MS. Heat intolerance seems, however, to be individually distributed among the MS patients, and may seem to be related to the degree of warmth.

Sixty patients with gait problems and without heat intolerance were included in a cross-over study. They were randomized to a 4-week inpatient physiotherapy based on the Bobath concept in Norway or Spain, with cross-over the year after. Data from five physical performance measures and six self-reported measures were collected at screening, baseline, after treatment and three and six months after both treatment-periods. Change over time within groups and comparisons of change between groups were analyzed by mixed models.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 60 years of age (both included).
* Multiple sclerosis according to the McDonald criteria
* Disability equivalent to Expanded Disability Status Score (EDSS) between 4.0 and 6.5 (both included)
* Prepared to and considered able to follow the protocol and to attend the planned visits during the whole study period.
* Given written informed consent

Exclusion Criteria:

* An active MS (attack or progression) during one month prior to inclusion or start of treatment.
* Received treatment with glucocorticoids the last month prior to inclusion or start of treatment.
* Excessive fatigue or severe cognitive dysfunction related to MS that would preclude safe participation in the protocol.
* Suffered from major depression or any other psychiatric disorder that would preclude safe participation in the protocol.
* Heat intolerance.
* Other serious concomitant disease that could preclude safe participation in the protocol.
* Alcohol or drug abuse or consumption that could preclude participation according to the protocol and to attend the planned visits during the whole study period.
* Breastfeeding or pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2006-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
6-minute walk test | 2 years

SECONDARY OUTCOMES:
Timed Up&Go | 2 years
10-metre timed walk | 2
Berg Balance Scale | 2
Trunk Impairment Scale | 2
Borg's Rating of Perceived Exertion | 2
Multiple Sclerosis Impact Scale (MSIS-29) | 2
Fatigue Severity Scale | 2
Numerical Rating Scale; gait, balance, pain | 2
Modified Health Assessment Questionnaire | 2
Patient Global Impression of Change | 2

CONTACTS AND LOCATIONS:
Overall Officials: Tori Smedal, MSc, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway